CLINICAL TRIAL: NCT03251365
Title: Intrabdominal Hyperthermic Chemotherapy Using Gemcitabine to Treat Pancreatic Carcinomatosis
Brief Title: Intrabdominal Hyperthermic Chemotherapy and Pancreatic Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General de Ciudad Real (Other)
Responsible Party: Principal Investigator, David Padilla-Valverde, Chief of Hepatobiliary Unit, Department of Surgery,HGUCR.Coordinator of Research Traslational Unit,HGUCR.Professor of Surgery, Faculty of Medicine, UCLM, Ciudad Real, Spain, Hospital General de Ciudad Real
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pancreathipec 1.0; 2016-004298-41 (EudraCT Number)
Record Dates: First submitted 2017-08-06; First posted 2017-08-16 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Resectable Pancreatic Adenocarcinoma
Keywords: Pancreatic cancer; Gemcitabine; Pancreatic carcinomatosis; Intrabdominal hyperthermic chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Characteristics of the Trial: This is a randomized,interventional, multidisciplinary study,phase II-III, involving several Services as General Surgery, Pathology, Oncology, Pharmacy, Gastroenterology and Radiology at the University General Hospital of Ciudad Real and the Faculty of Medicine, and Translational Research Unit,HGUCR.The study is opened to the incorporation of other centers that increase the power of the obtained results.
Who Masked: Participant, Investigator
Masking Description: After explaining the treatment to develop once informed of the characteristics of pancreatic cancer to the patient, we will explain in detail the clinical trial that we are going to develop. After obtaining the informed consent, authors will start the randomly distribution of patients A list of randomization to 42 patients will be developed by a computer program that simulates the extraction procedure of numbered balls and the correlative allocation to each of the codes.
  Randomization is by block, thereby ensuring a balanced number of subjects per treatment. Then a scrambling code in which randomly assigned treatment to each code will be developed.
  The randomization code and study randomization list shall be kept only for the person that will carry the allocation of treatments.Randomization of patients will be performed centrally. Each patient is assigned to a sequential number of the centralized list of inclusion and appropriate treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I, Normal (No Intervention): Group I. After cytoreductive surgery, R0, and intestinal reconstruction, the patient after multidisciplinary study will receive adjuvant treatment with iv gemcitabine , 1000 mg / m2 for at least 4 cycles
- Group II,experimental.HIPEC-Gemcitabine (Experimental): • Group II.After a R0 cytoreductive surgery, HIPEC is performed with gemcitabine, 120mg / m2 for 30' + adjuvant treatment with iv gemcitabine , 1000 mg / m2 for at least 4 cycles
  Interventions: Drug: HIPEC-gemcitabine

INTERVENTIONS:
Drug: HIPEC-gemcitabine — • Group II.After a R0 cytoreductive surgery, HIPEC is performed with gemcitabine, 120mg / m2 for 30' + adjuvant treatment with iv gemcitabine , 1000 mg / m2 for at least 4 cycles
  Arms: Group II,experimental.HIPEC-Gemcitabine

SUMMARY:
A randomized, multidisciplinary study, Phase II-III clinical trial.The study is opened to the incorporation of other centers that would increase the power of the obtained results . Our hypothesis considers that using Hyperthermic Intra-abdominal Chemotherapy,HIPEC, with gemcitabine after cytoreductive surgery ,will decrease tumor progression of pancreatic cancer by reducing the neoplastic volume and subpopulation of pancreatic cancer stem cells, improving the survival of patients with pancreatic cancer, and decreasing the recurrence of the disease

DETAILED DESCRIPTION:
According to the incidence in the area of the University General Hospital, Ciudad Real, HGUCR, authors will include a population of 42 patients, n = 21 in each group, I and II, with diagnosis of adenocarcinoma of the pancreas, which will be surgically resected with curative intention, in the next two years, 2017-2018, with extended follow-up for at least two years more for survival study Accepting an alpha risk of 0.05 and a beta risk of 0.2 in a bilateral contrast, 21 subjects were required in the first group and 21 participants in the second Group to detect as statistically significant difference between two proportions, for group I is expected to be 0.05 and for Group II 0.4, in relation to survival in five years. It has been estimated a rate of loss of patients of 10%

* Group I. After cytoreductive surgery, R0, and intestinal reconstruction, the patient after multidisciplinary study will receive adjuvant treatment with iv gemcitabine , 1000 mg / m2 for at least 4 cycles
* Group II.After a R0 cytoreductive surgery, HIPEC is performed with gemcitabine, 120mg / m2 for 30' + adjuvant treatment with iv gemcitabine , 1000 mg / m2 for at least 4 cycles The aim is identifying morbidity and mortality associated to treatment by cytoreductive surgery and HIPEC with gemcitabine+ systemic chemotherapy,Group II, respect to a conventional treatment group that includes cytoreductive surgery with systemic chemotherapy, Group I,and identifying survival of the experimental Group with treatment with cytoreductive surgery and HIPEC with gemcitabine ,respect to the conventional treatment group,GI

ELIGIBILITY:
Inclusion Criteria:

· Resectable pancreatic adenocarcinoma

Exclusion Criteria:

* Voluntary refusal to participate in the trial
* Existence of distant disease that contraindicates the surgical treatment
* Patients with preoperative or intraoperative locoregional unresectable pancreatic cancer
* Existence of synchronous neoplastic disease
* Exclusion after perioperative anesthetic study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2017-07-27 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Morbidity | 30 days
  • Identify morbidity associated to treatment by cytoreductive surgery and HIPEC with gemcitabine+ systemic chemotherapy,Group II, respect to a conventional treatment group that includes cytoreductive surgery with systemic chemotherapy, Group I
Survival | 18 months
  • Identify survival of the experimental Group with treatment with cytoreductive surgery and HIPEC with gemcitabine ,respect to the conventional treatment group,GI

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Ciudad Real, HGUCR, Ciudad Real, Spain

IPD SHARING:
Plan to Share IPD: Undecided